CLINICAL TRIAL: NCT00955396
Title: A Randomized, Double-blind, Placebo-controlled Cross-over Study to Investigate the Effect of GSK1014802 on Ambulatory Blood Pressure
Brief Title: Study to Investigate the Effect of GSK1014802 on Ambulatory Blood Pressure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 113210; SCB113210
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteer
Keywords: sodium channel blocker; ambulatory blood pressure
MeSH Terms: interventions — vixotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Period 1 (Other)
  Interventions: Drug: GSK1014802; Drug: Placebo
- Period 2 (Other)
  Interventions: Drug: GSK1014802; Drug: Placebo

INTERVENTIONS:
Drug: GSK1014802 — Tablets
  Other Names: BIIB074 and CNV1014802
Drug: Placebo — Tablets

SUMMARY:
In this study the investigators will determine whether there is any effect of GSK1014802 on ambulatory blood pressure. This will be a randomized, double-blind, placebo-controlled, repeat dose, 2 period cross-over study conducted in healthy male and female subjects. Approximately 60 subjects will be randomised to receive GSK1014802 400 mg bid and placebo for 36 days with at least 1 week between treatment sessions. A follow-up will occur 7-14 days after the last dose.

DETAILED DESCRIPTION:
This study, previously posted by GlaxoSmithKline (GSK), was transitioned to Convergence Pharmaceuticals, Ltd., which spun off from GSK. Convergence Pharmaceuticals, Ltd., has now been acquired by Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests, liver function and cardiac monitoring.
* A female subject is eligible to participate if she is of:

Non-childbearing potential Child-bearing potential and agrees to use a contraception method.

* Male subjects must agree to use a contraception methods
* Body weight ≥ 50 kg and BMI within the range 19 - 40.0 kg/m2 (inclusive).
* Arm circumference ≥ 24 and ≤ 42 cm at mid level.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug screen.
* Alcohol levels above the legal limit for driving at screening and the detection of any alcohol within 24 h prior to the start of dosing in Treatment Periods 1 and 2.
* A positive test for HIV antibody.
* History of regular excessive alcohol consumption within 6 months of the study
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including any antihypertensive agent including diuretics, vitamins, herbal and dietary supplements
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Subjects who work at night or whose work schedule includes rotating night time (10:00 PM to 6:00 AM) work.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Average daily caffeine intake equivalent to > 4 cups of coffee or > 6 cups of tea.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Consumption of aged cheeses and meats, soy sauce and other tyramine rich sources within 1 day prior to the baseline assessments.
* Current or past history of symptomatic orthostatic hypotension or history of unexplained vasovagal episode(s).
* History of known or suspected seizures, including infantile febrile, unexplained significant and recent loss of consciousness or history of significant head trauma with loss of consciousness or a family history (first degree relative) of epilepsy or seizures (fits).
* Any history of suicidal behaviour or suicidal ideation of type 4 or 5 on the C-SSRS within 3 months of the screening visit.
* History or currently diagnosed sleep apnea.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07-31 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
Change in 24 h average SBP and DBP from Baseline to Day 36. | 36 days

SECONDARY OUTCOMES:
Change in 24 h average SBP and DBP from Baseline to Day 15. Change in average SBP and DBP within a dosing interval (12 h) from Baseline to Days 14 and 35. | 35 days
Change in 24 h average SBP and DBP from Baseline to Days 15 and 36 in subjects with baseline SBP 120-139 mmHg and also DBP 80-89 mmHg. | 36 days
Change in day-time outpatient (6:00 AM to 10:00 PM) SBP and DBP from Baseline to Days 15 and 36. | 36 days
Change in night-time outpatient (10:00 PM to 6:00 AM) SBP and DBP from Baseline to Days 15 and 36. | 36 days
Change in 24 h average ambulatory heart rate from Baseline to Days 15 and 36. | 36 days
Proportion of patients whose 24 h systolic and diastolic BP increased by < 5, 5-9, 1014, 15-19, and > 20 mm Hg compared to baseline. | 36 days
PK parameters of GSK1014802 following a single oral dose of GSK1014802 to healthy female subjects: Cmax, tmax, AUC (0-t) and, if possible, AUC(0-∞), λz and terminal phase half-life to healthy female subjects. | 1 day
PK parameters of GSK1014802 following repeated oral doses of GSK1014802 given twice daily to healthy male and female subjects: Cmax, tmax, AUC(0-12). | 36 days
PK/PD analyses to examine the correlation between ambulatory blood pressure and plasma levels and/or metrics of the systemic exposure (Cmax, AUC) of GSK1014802. | 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Medical Director, Study Director — Biogen
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States